CLINICAL TRIAL: NCT05550051
Title: Lignocaine Nebulization Versus Airway Block for Awake Nasal Fiberoptic Intubation in Patients With Head and Neck Burns. A Randomized Controlled Study.
Brief Title: Lignocaine Nebulization Versus Airway Block for Awake Nasal Fiberoptic Intubation in Patients With Head and Neck Burns.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sameh Refaat, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R121/2022
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Practicality, Efficacy, and Ease of Lignocaine Nebulization Compared to Traditional Upper Airway Block for Awake Nasal Fiberoptic Intubation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lignocaine nebulization before awake nasal fiberoptic intubation (Active Comparator): Patients will have lignocaine nebulization by using 3 ml of lignocaine 2%, with O2 flow rate 10 l/min to deliver 60 mg lignocaine, of which about 25% is absorbed, and patients were encouraged to inhale deeply to facilitate further delivery of the anesthetic in their airway. After finishing the nebulization setting the patient will be asked about facial, nasal, and oral numbness if no numbness, the patient will have another nebulization setting.
  Interventions: Procedure: Awake nasal fiberoptic intubation
- Upper airway block before awake nasal fiberoptic intubation (Active Comparator): Upper airway block by using about lignocaine 2%, the block will be performed by:
  1. Bilateral superior laryngeal nerve block and will be performed by slight neck extension to identify the hyoid bone. Insert the needle laterally aiming at the greater cornu, and after hitting the bone, it will slide inferiorly, and 2 mL of 2% lignocaine will be injected blocking both the internal and the external branches of the superior laryngeal nerve.
  2. Trans tracheal instillation for recurrent laryngeal nerve block and will be performed by extending the neck to identify the midline and palpate the cricoid cartilage. The cricothyroid membrane lies above the cricoid cartilage. A needle will be inserted in the cricothyroid membrane while aspirating and once air bubbles appears, 5ml of 4% lignocaine will be injected resulting in cough and dispersing of the LA, blocking the nerve.
  Interventions: Procedure: Awake nasal fiberoptic intubation

INTERVENTIONS:
Procedure: Awake nasal fiberoptic intubation — Lignocaine nebulization for upper airway block during awake nasal fiberoptic intubation

SUMMARY:
This study evaluates the efficacy and ease of lignocaine nebulization to deliver anesthesia to the upper airway of patients with head and neck burns undergoing reconstructive surgery in need of awake nasal fiberoptic intubation compared to the traditional upper airway nerve block.

DETAILED DESCRIPTION:
Adequate preparation for Awake Fiberoptic Intubation (AFOI) is an art of anesthesia which includes, many methods such as blocking nerves supplying the upper airway including the superior laryngeal, recurrent laryngeal, and glossopharyngeal nerves. Topical anesthesia via a special cannula as you proceed, and lignocaine nebulization. Succeeding in blocking the airway adequately is the first step towards a successful AFOI.

Although many studies have been done to compare the topical anesthesia technique versus the airway block techniques but theses studies have ignored the fact that in many cases of difficult airway indicated for AFOI there is limited or even absent neck mobility, and mouth opening both which are mandatory to perform an adequate airway neural block.

After anesthetizing the airway in both groups either by nebulization or airway block, an anesthesiologist who will be blinded to the study groups will perform the (AFOI) by using an endotracheal tube size 7.5 mm internal diameter endotracheal tube for males and 7 mm for female patients.

Vital signs such as HR, BP, and oxygen saturation (SpO2) will be recorded recorded immediately after intubation and 5 min postintubation and at every 10 minutes during surgery.

The patient response, and satisfaction with the technique will be recorded by using the revised non verbal pain scale (NVPS-R).

The (NVPS-R) is a multidimensional instrument formed of three behavioral (face, activity/movement, and guarding) responses, physiological indicators, and RR.

Patients will be randomly divided into two groups using a computer generated random number chart. Group (AB) will undergo AFOI after performing an airway block prior to the procedure while group (LN) will undergo AFOI after lignocaine nebulization 30 minutes prior to the procedure.

Group (AB) will have an upper airway block by using about lignocaine 2%; the following nerves will be blocked.

Bilateral superior laryngeal nerve block and will be performed after placing the patients in a supine position, with slight neck extension to identify the hyoid bone. Sterilization of the site of injection by 10% povidone iodine will be performed. After identification of the hyoid bone the bone will be move towards the site of injection, where a sterile 25G needle will be inserted laterally aiming at the greater cornu, and after hitting the bone with the needle, it will slide under the bone inferiorly, and 2 mL of 2% lignocaine will be injected blocking both the internal and the external branches of the superior laryngeal nerve.

Trans tracheal instillation for recurrent laryngeal nerve block and will be performed by placing the patient supine, with the neck extended to identify the midline and palpate the cricoid cartilage. The cricothyroid membrane lies above the cricoid cartilage. A 22G needle will be inserted perpendicular to the cricothyroid membrane to penetrate it while aspirating and once air bubbles appear this will mean that we are intra tracheal, then injection of 5ml of 4% lignocaine will result in coughing and dispersing of the LA, blocking the nerve.

While patients in group (LN) will have lignocaine nebulization by using 3 ml of lignocaine 2%, with O2 flow rate 10 l/min to deliver 60 mg lignocaine, of which about 25% is absorbed, and patients were encouraged to inhale deeply to facilitate further delivery of the anesthetic in their airway. After finishing the nebulization setting the patient will be asked about facial, nasal, and oral numbness if no numbness, the patient will have another nebulization setting.

ELIGIBILITY:
Inclusion Criteria:

* All patients above 18 years with ASA classification II, III, and no known hypersensitivity for local anesthetics

Exclusion Criteria:

* Patient refusal
* Patients under 18 years
* Patients suffering from coagulopathies or bleeding tendencies
* Patients with ASA 4 classification
* Non cooperative patients
* Patients undergoing extensive facial reconstruction
* Patients with known hypersensitivity to lignocaine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
Patient comfort during performing awake nasal fiberoptic intubation | 5 minutes
  Will be measured by the revised non verbal pain sale
Time to performing awake nasal fiberoptic intubation | 5 minutes
  Will be measured by calculating the time to awake nasal fiberoptic intubation

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Refaat, MD, Principal Investigator — Ain Shams University
Locations (1):
- Sameh Refaat, Cairo, Egypt